CLINICAL TRIAL: NCT07047911
Title: Predictors of Morbidity in Perforation Peritonitis: A Prospective Observational Study From a Tertiary Care Centre in North India
Acronym: PERIMOPP
Status: Completed | Type: Observational
Sponsor: Government Medical College, Patiala (Other Government)
Responsible Party: Principal Investigator, Lakshay Singla, Doctor, Government Medical College, Patiala
Other Study IDs: GMC-PERITONITIS-2016
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Peritonitis Infectious, Gastrointestinal Perforation, Surgical Infection, Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational only - surgical management not assigned by study — Observational only - surgical management not assigned by study

SUMMARY:
This is a prospective observational cohort study conducted at a tertiary care hospital in North India. The study aims to evaluate clinical and biochemical predictors of postoperative morbidity in patients undergoing emergency laparotomy for gastrointestinal perforation peritonitis. Data on patient demographics, comorbidities, surgical timing, renal function, and complications were collected and analyzed to identify factors associated with increased morbidity. The findings are expected to support early risk stratification and improved clinical management of surgical emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) with gastrointestinal perforation-induced peritonitis

Exclusion Criteria:

* Primary peritonitis, anastomotic leaks, refusal of surgery, or patients discharged against medical advice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 adult patients were enrolled prospectively over a 2-year period at Government Medical College & Rajindra Hospital, Patiala.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-03-10 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
Post operative morbidity | 30days
Post operative morbidity | 30 days